CLINICAL TRIAL: NCT05700123
Title: Non-pharmacological Methods for the Control of Anxiety and Pain During Outpatient Hysteroscopy (Metodiche Non Farmacologiche Per il Controllo di Ansia e Dolore Durante Isteroscopia Ambulatoriale)
Brief Title: Non-pharmacological Methods for the Control of Anxiety and Pain During Outpatient Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Gaetano Riemma, Principal Investigator, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0013700/i
Record Dates: First submitted 2023-01-13; First posted 2023-01-26 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Video (Experimental)
  Interventions: Procedure: In-Office Hysteroscopy
- Music (Experimental)
  Interventions: Procedure: In-Office Hysteroscopy
- Vocal-Local (Active Comparator)
  Interventions: Procedure: In-Office Hysteroscopy

INTERVENTIONS:
Procedure: In-Office Hysteroscopy — In-office hysteroscopic procedures were conducted using a 5mm continuous flow Office Hysteroscope using a vaginoscopic, no-touch, approach

SUMMARY:
The administration of pharmacological and non-pharmacological aids during in-office hysteroscopic surgery is often used to both relieve the patient from discomfort and facilitate the operator in performing the procedure. The investigators aim to test the hypothesis that watching a video clip or listening to music would act as non-pharmacological relief for reducing anxiety and pain during in-office hysteroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal and postmenopausal women
* Indication for in-office operative hysteroscopy

Exclusion Criteria:

* Denied consent
* Use of analgesic drugs before the procedure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
The anxiety, evaluated by means of State-Trait Anxiety Inventory (STAI) questionaries | 24 hours
  20 (better) - 80 (worse)
post-hysteroscopic pain, evaluated using a 1-10 Numeric Rating Scale (NRS) | 24 hours
  1 (better) - 10 (worse)

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Franciscis, MD PhD, Study Chair — Università della Campania Luigi Vanvitelli; Gaetano Riemma, Principal Investigator — Università della Campania Luigi Vanvitelli
Locations (3):
- Italy (3):
  - University of Bari, Bari
  - University of Cagliari, Cagliari
  - University of Campania "Luigi Vanvitelli", Napoli

IPD SHARING:
Plan to Share IPD: No